CLINICAL TRIAL: NCT05641389
Title: Improving Remote Breathalyzer Procedures Used by Clinicians and Researchers to Remotely Monitor Alcohol Use
Status: Recruiting | Type: Observational
Sponsor: University of North Texas, Denton, TX (Other)
Collaborators: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Donald Dougherty, Department Chair, University of North Texas, Denton, TX
Other Study IDs: 22-173
Record Dates: First submitted 2022-11-15; First posted 2022-12-07 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Alcohol Monitoring; Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Monitoring Group: Participants will be monitored via a transdermal monitor for four weeks. They will give four breath samples a day for these weeks as well as 5 Blood spot samples.
  Interventions: Other: Monitoring

INTERVENTIONS:
Other: Monitoring — Participants will be monitored for alcohol use.

SUMMARY:
Remote breath alcohol monitors have been increasingly adopted for use in clinical, research and forensic settings to monitor alcohol use because they offer several key advantages over other available monitoring methods. However, it remains unknown if remote breathalyzers reliably detect alcohol use because there is up to a 10-hour window of time when breath samples are not obtained (to allow for sleeping). Additionally, the investigators will examine whether a supplemental measurement of a blood alcohol use biomarker (phosphatidylethanol) can confirm abstinence and/or detect individuals engaging in late-evening drinking to avoid the negative consequences associated with detected alcohol use.

DETAILED DESCRIPTION:
Devices that can continuously and/or remotely monitor alcohol use have created new opportunities for both research and intervention, initially with transdermal alcohol monitors (TAMs) that continuously and remotely detect alcohol excreted through the skin. TAMs were first designed and used in the criminal justice system, but their disadvantages have limited widespread adoption (e.g., availability, cost, size, interference with physical activities, and stigma) (Allessi et al., 2017; Caluzzi et al., 2019). Thus, other alcohol monitoring technologies (and procedures) to detect and characterize alcohol consumption are being developed and used. One example is remote breathalyzers (e.g., SCRAM Remote Breath®), a potential alternative to TAMs. They are small, can be used daily and more privately, use Automated Facial Intelligence™ (AFI™) technology to verify identity, and have safeguards to prevent circumvention (SCRAM, 2020). Heavy drinking may go undetected when using prescribed remote breathalyzer monitoring protocols. Remote breathalyzers are being used more frequently in legal and clinical research settings (e.g., Alessi & Petry, 2013; Koffarnus et al., 2018; Moody et al., 2018; Nehlin et al., 2018; Recovery Healthcare Corporation, personal communication, June 22, 2021; Skipper et al., 2014). The underlying assumption is that breathalyzers objectively detect alcohol consumption. In fact, among social drinkers (n = 12), remote breath alcohol concentration (BrAC) monitoring protocols had a 98.8% rate of correspondence with self-reported drinking (Skipper et al., 2014), where there were no drinking-associated contingencies/consequences. Manufacturer monitoring protocols have not been validated among individuals who do have contingencies/ consequences associated with detected drinking. Remote breath sampling protocols may provide ample opportunity for individuals to drink heavily, especially among populations where detected drinking is associated with penalties. Importantly, when contingencies are present, individuals may adopt or adjust their drinking patterns to "beat" the system. For instance, procedures used in the judicial system (which correspond with manufacturer recommendations), individuals are prompted to submit 4 breath samples/day, beginning at a start time chosen by the person being monitored and then every 5 hours thereafter (e.g., 7am, 12pm, 5pm, 10pm). Each person's schedule for sampling is the same every day and breath samples must be submitted within an hour after prompting. Therefore, these schedules have "on- and off-cycle" times, with the on-cycle schedule covering only ~15 hours of each day. The off-cycle schedule, from the submission of the last sample on one day to the first sample the next day, allows time for sleep, but during this time (up to 10 hours, including an allowance for the sampling window) drinking could occur. People could drink right after their last breath sample (e.g., 10pm) and still submit a negative BrAC (<.02 g/dL) the next day (required by 8am). BrAC ≥.02 g/dL are considered positive for alcohol use (NHTSA, 2018). Based on our prior alcohol self-administration study, at varying levels of intoxication, both men and women could be below .02 g/dL within ~6 hours (Figure 1; Hill-Kapturczak et al., 2015), showing considerable latitude for engaging in drinking and not violating monitoring criteria. Thus, it is unknown if remote BrAC monitors can yield reliable and valid measures of drinking events in those who: (a) may find it difficult to control drinking, and (b) are motivated to avoid detection of drinking due to consequences.

ELIGIBILITY:
Inclusion Criteria:

•≥ 21 years of age

•Either convicted of a DWI offense in the past 2 years but not court-mandated to undergo continuous alcohol monitoring or reporting driving while intoxicated in the past year or report ≥ 10 heavy drinking episodes during the past month (heavy drinking episodes count as more than 3 drinks in a day for females and 4 or more alcoholic drinks in a day in a male).

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study population is consisted of members of the DFW metroplex.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Transdermal Alcohol Content | They will be placed on the device starting at the first visit and wear it for four weeks till the last visit.
  Measurement produced while wearing Transdermal Alcohol Monitor
Measurement of Phosphatidylethanol | Once every week for four weeks.
  Measuring Phosphatidylethanol via blood spot cards. THis is a measurement of alcohol use.

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Texas, Denton, Texas, United States